CLINICAL TRIAL: NCT05277298
Title: A Prospective Household Study of SARS-CoV-2, Influenza, and Respiratory Syncytial Virus Community Burden, Transmission Dynamics and Viral Interaction in South Africa (the PHIRST-C Study)
Brief Title: Household Study of COVID-19, Influenza and RSV Burden, Transmission Dynamics and Viral Interaction in South Africa
Acronym: PHIRST-C
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Institute for Communicable Diseases, South Africa (Other)
Collaborators: Perinatal HIV Research Unit of the University of the Witswatersrand (Other); University of Witwatersrand, South Africa (Other); Centers for Disease Control and Prevention (U.S. Federal Agency); Institute for Scientific Interchange, Torino, Italy (Unknown); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Other Study IDs: PHIRST-C
Record Dates: First submitted 2020-12-30; First posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: SARS-CoV-2 Infection; Influenza; Respiratory Syncytial Virus (RSV)
Keywords: SARS-CoV-2; influenza; RSV; household transmission; COVID-19
MeSH Terms: conditions — COVID-19; Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Respiratory samples (nasal swab), serological samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to characterize the community burden (including the clinical features) and transmissibility of SARS-CoV-2 within the context of a functional antibody response. In addition,the study will assess the effect of the interaction of SARS-CoV-2 with influenza virus and RSV on disease severity and transmission dynamics. A household-level prospective cohort study will be conducted in one rural and one urban community located in Mpumalanga Province and North West Province, respectively. The study will be conducted for 12 months of intensive follow up (July 2020 to August 2021) with a post-intensive follow-up continuing for a further 16 months (until December 2022). Two hundred households; 1,000 study participants of all ages; will be randomly selected from a list of 327 hoseholds that participated and successfully completed a 10-months follow-up period in a study similar to that currently proposed, but directed at community burden and transmission dynamics of influenza, respiratory syncytial virus and other respiratory pathogens. Each household and household member will be enumerated and the HIV infection status and the level of immunosuppression of HIV-infected individuals will be assessed. Each household member will be followed twice per week during the intense follow-up period (12 months) of the study. During this period upper respiratory tract samples will be collected irrespective of presence of symptoms and data on key symptoms, healthcare seeking, hospitalization and death will be captured at each follow up visit. Respiratory samples will be tested by reverse transcriptase real-time polymerase chain reaction (rRT-PCR) for SARS-CoV-2, influenza and RSV, and selected samples will be cultured and sequenced. An infection risk questionnaire will be administered to all study participants at enrollment and every month thereafter. Sera will be collected at enrollment and every 2 months during the 12-month intense follow-up period from all participants. In addition, sera will be collected every 2 months for a further 6 months following the 12-month intense follow-up period from study participants that tested positive for SARS-CoV-2 by rRT-PCR on respiratory specimens at 14, 16 and 18 months and from all study participants at 18 months. Sera will be tested for the presence of SARS-CoV-2, influenza and RSV antibodies. Wearable proximity sensors will be deployed for 8-12 days in each household over the 6-month intense follow-up period.

DETAILED DESCRIPTION:
Background and justification: On 31 December 2019, the World Health Organization (WHO) was alerted to a cluster of pneumonia cases of unknown etiology in patients in Wuhan City, Hubei Province of China, which, one week later, was attributed to a novel coronavirus (severe acute respiratory syndrome coronavirus 2: SARS-CoV-2). Given its rapid spread globally, WHO declared that the outbreak of SARS-CoV-2 met pandemic criteria on 11th March 2020. By mid-April 2020 more than 2.5 million cases and more than 170,000 deaths have been laboratory-confirmed in 210 countries and territories.

Influenza virus is responsible for elevated morbidity and mortality globally every year. In South Africa annual seasonal influenza epidemics occur during the winter months (May-October, with peak transmission in June-July) and result in an estimated 19 million symptomatic infections, 128,000 severe cases and 11,000 deaths on average every year.

Human respiratory syncytial virus (RSV) is the commonest cause of childhood acute lower respiratory tract infection, especially among infants <3 months of age. In South Africa RSV circulates throughout the year with peak transmission occurring usually during February-April. Nonetheless, from systematic virologic surveillance data delayed RSV transmission is expected to occur in South Africa in 2020. This has the potential to result in concomitant SARS-CoV-2, influenza and RSV peak transmission in the country.

HIV incidence remains high in South Africa. Similarly, rates of pulmonary tuberculosis (PTB), with concomitant damage to lung tissue, remain persistently high despite concerted national efforts. HIV and PTB infections have been associated with an increased risk of severe illness (i.e., hospitalization and death) following infection with common respiratory pathogens, including influenza and RSV, even among individuals on antiretroviral therapy.

Understanding the community burden, transmissibility potential and clinical features of illness associated with SARS-CoV-2 infection is critical to inform the design and duration of containment and mitigation measures, both locally and globally. An accurate estimation of risk factors for community transmission, acquisition and duration of infectiousness is crucial to inform guidance for public health measures to limit transmission as well as models for epidemic forecasting for this and potential future epidemics. Moreover, factors specific to South and sub-Saharan Africa (SSA) such as HIV, tuberculosis, high proportion of the population who are children, malnutrition, and limited healthcare resources have the potential to impact both the transmission dynamics, progression and prognosis of SARS-CoV-2 disease; as well as the burden on the healthcare system and society.

Whereas knowledge has been gained on the transmissibility and clinical features of SARS-CoV-2 since its emergence several key questions related to the natural history of the virus remain poorly answered, notably in African context. In particular, the community attack rate by age, the role of children in community and household transmission, the asymptomatic infected fraction, the role of asymptomatic individuals in transmission, the interaction of SARS-CoV-2 with other common respiratory pathogens such as influenza and RSV, the risk of reinfection with SARS-CoV-2 and the correlation between PCR-confirmed infection and serologic response among others, remain poorly understood. Critically, the effect of HIV infection on transmission and disease severity associated with SARS-CoV-2 infection is unknown. South Africa has an HIV prevalence of approximately 15% in the general population, representing over 7 million people of whom over 5 million are taking antiretroviral therapy.

Aim: In urban and rural South African environments, the study aims to characterize the community burden (including the clinical features) and transmissibility of SARS-CoV-2 within the context of a functional antibody response. In addition, the effect of the interaction of SARS-CoV-2 with influenza virus and RSV on disease severity and transmission dynamics will be assessed. This will be undertaken from an early stage throughout the epidemic in South Africa.

Primary objectives:

1. To estimate the community burden of SARS-CoV-2, including:

   1.1 the incidence of SARS-CoV-2 infection in the community as determined by polymerase chain reaction (PCR) and serologic assays; 1.2 the correlation between individuals that seroconverted for SARS-CoV-2 and tested positive by PCR; 1.3 the incubation period and the symptomatic fraction associated with SARS-CoV-2 infection; 1.4 the spectrum of severity associated with symptomatic infections; 1.5 the fraction of individuals with symptomatic infection seeking medical care; and 1.6 the effect of the interaction of SARS-CoV-2 with influenza and RSV on disease severity.
2. To assess the transmission dynamics of SARS-CoV-2 infections in the community, including:

2.1 the estimation of the SARS-CoV-2 household secondary infection risk (SIR), generation time and length of shedding; 2.2 the estimation of the probability of transmission of SARS-CoV-2 infection between individuals (both symptomatic and asymptomatic/presymptomatic) within the household and potentially the community; 2.3 the estimation of the SARS-CoV-2 effective reproduction number (Rt) and its variation over time in the community; and 2.4 the effect of the interaction of SARS-CoV-2 with influenza and RSV on transmission dynamics.

Methods: A household-level prospective cohort study will be conducted in one rural and one urban community located in Mpumalanga Province (the Agincourt demographic surveillance site) and North West Province (Klerksdorp), respectively. The study will be conducted for 14 months of intensive follow up (July 2020 to August 2021) with a post-intensive follow-up continuing for a further 16 months (until December 2022).

Two hundred households; 100 per site with expected average number of household members of 5 resulting in 1,000 study participants of all ages; will be randomly selected from a list of 327 households that participated and successfully completed a 10-months follow-up period in a study similar to that currently proposed, but directed at community burden and transmission dynamics of influenza, respiratory syncytial virus and other respiratory pathogens (the PHIRST study conducted during 2016-2018 in the same two communities). The approached households will be re-assessed for study eligibility (i.e., a minimum of 3 household members and at least 80% of household members consenting to participate). The households in the 2016-2018 PHIRST study were identified by randomly selected geo-coordinates within the two communities. Baseline characteristics for this cohort are already available and will be re-ascertained after obtaining consent. Consenting household members that have entered the household since termination of the 2016-2018 PHIRST study will be also enrolled. Each household and household member will be enumerated and the HIV infection status and the level of immunosuppression of HIV-infected individuals will be assessed (if unknown) in consenting individuals.

Each household member will be followed twice per week during the intense follow-up period (12 months) of the study. During this period upper respiratory tract samples will be collected irrespective of presence of symptoms and data on key symptoms, healthcare seeking, hospitalization and death will be captured at each follow up visit on a REDCap tablet-based real-time database. Respiratory samples will be tested by reverse transcriptase real-time polymerase chain reaction (rRT-PCR) for SARS-CoV-2, influenza and RSV, and selected samples will be cultured and sequenced. An infection risk questionnaire will be administered to all study participants at enrollment and every month thereafter. Sera will be collected at enrollment and every 2 months during the 12-month intense follow-up period from all participants. In addition, sera will be collected every 2 months for a further 6 months following the 12-month intense follow-up period from study participants that tested positive for SARS-CoV-2 by rRT-PCR on respiratory specimens at 14, 16 and 18 months and from all study participants at 18 months. Sera will be tested for the presence of SARS-CoV-2, influenza and RSV antibodies. Wearable proximity sensors will be deployed for 8-12 days in each household over the 6-month intense follow-up period.

Impact: This study will provide essential information on the natural history of the virus that will impact decisions on optimal strategies for the containment and mitigation of the current and potential future epidemics of SARS-CoV-2 locally, regionally and globally.

ELIGIBILITY:
Inclusion Criteria:

* Households/individuals that consent to participate to the study; and that are planning to reside in the selected community for the duration of the study.
* Provide at least one serum sample in the intensive follow up period, for individuals five years and older and
* Households should have at least 3 or more.

Exclusion Criteria:

Households that:

* Non-eligible households will be households that were not randomly selected, that were selected but did not consent to participate to the study or, that have >20% of household members who do not consent for inclusion in the study.

Ages: 0 Days to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Mpumalanga Province site
  The population is approximately 120,000 people living in 20,000 households While HIV prevalence is high, life expectancy is improving with marked epidemiological transition leading to rising prevalence of non-communicable disease including cardio-metabolic conditions and stroke.
  North West Province Site
  Klerksdorp is located in the local municipality of Matlosana in North West Province and has a population of over 385,000 people and is 115 km2. The townships are organized into extensions that include mostly single-family houses and shacks. Prevalence of HIV in Klerksdorp is approximately 12%.
Sampling Method: Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Describe the symptomatic fraction of SARS-CoV-2 infections among individuals in household cohort in an rural and urban setting, South Africa 2020/2021. | 14 months
  The proportion of SARS-CoV2 infection that are symptomatic. This will be stratified by age, underlying conditions, HIV infection.
Describe the household secondary infection risk of SARS-CoV-2 infection among individuals in a household cohort in an rural and urban setting, South Africa 2020/2021. | 14 months
  The number of secondary cases in a household divided by the total number of susceptible gives the secondary attack risk during the 14months of follow-up. This will be explored by underlying conditions, age and HIV status
Describe the serial interval for SARS-CoV-2 in households over 14 months of follow-up in an urban and rural setting, South Africa 2020/2021 | 14 months
  Calculate the time between successive cases in a each household as documented by onset of symptoms and/or PCR positive test.
Describe the duration of shedding of SARS-CoV-2 in a household cohort in an rural and urban setting, South Africa 2020/2021. | 14 month
  The duration of PCR positive SARS-CoV-2 infection in individual over 14 months of follow-up, including describing the interval by age, HIV status and underlying conditions.
Describe the incidence of infection by PCR and serology in a household cohort in a rural and urban setting, South Africa 2020/21 | 14 months
  The number of new cases of symptomatic illness recorded by symptoms reported cohort over the 14 months of follow-up. Including estimating a person time to follow-up incident rate
Describe the incidence illness by PCR and/or serology in a household cohort in a rural and urban setting, South Africa 2020/21 | 14 months
  Describe the incidence of infection by PCR and serology in a household cohort over 14 months of follow-up, in a rural and urban setting, South Africa 2020/21

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Kahn, MD, PhD, Principal Investigator — MRC/Wits Rural Public Health and Health Transitions Research Unit (Agincourt), Bushbuckridge, South Africa; Neil Martinson, MD, PhD, Principal Investigator — Perinatal HIV Research Unit, Johannesburg
Locations (2):
- South Africa (2):
  - MRC/Wits Rural Public Health and Health Transitions Research Unit (Agincourt), Bushbuckridge, South Africa, Agincourt, Mpumalanga
  - Perinatal HIV Research, Klerksdorp, North West

IPD SHARING:
Plan to Share IPD: Yes
The study investigators will update the study results to the clinicaltrials.gov site and publish interim results in peer review journals within 6 months of study start.
Supporting Information: Study Protocol, ICF
Time Frame: Protocol informed consent will be uploaded to PHIRST-C webpage by by 31/1/2021.
Access Criteria: open access, will be added once available
URL: https://www.nicd.ac.za/centres/centre-for-respiratory-disease-and-meningitis/